CLINICAL TRIAL: NCT05191511
Title: Assessment of Safety Distance of Far-Infrared Therapeutic Device to Human Skin
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Tainan Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Sponsor
Other Study IDs: 20180101
Record Dates: First submitted 2021-10-04; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-09

CONDITIONS: Far- Infrared Burn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Far- infrared — safety of far- infrared

SUMMARY:
Abstract The equipment "infrared therapeutic device" is widely used in various medical institutions in Taiwan. The infrared therapeutic device improves the blood circulation, relieves muscle stiffness and pain by the heat energy radiated by the infrared light, and has a significant relief effect on patients with joint pain, muscle soreness, and back discomfort. However, the principle of the infrared therapeutic device is thermal energy, and there is no complete literature on the parameters such as treatment intensity and time and the full distance. In addition, the literature on the damage that can be caused is not based on clinical evidence, and there is no standardization study on the use of equipment, so it is hoped that this test will explore the safety distance of infrared therapeutic devices.

The project is expected to recruit 50 people from 20 years old to 75 years old in the Chinese Medicine Clinic of Tainan Hospital of the Ministry of Health and Welfare, which is included in the diagnosis of osteoarthritis, degenerative arthritis, osteoporosis and other related Chinese medicine clinics. In patients with diseases, the main complaint must include patients with lower back pain and back pain. Subjects should exclude diseases that may be affected by chemoradiotherapy, cardiovascular disease, anemia, hypertension, etc., and exclude dermatitis, skin irritation, and erythema. Skin diseases such as lupus. The test site is the TCM clinic of Tainan Hospital of the Ministry of Health and Welfare. The air conditioner is fixed at a constant temperature of 28 degrees. The output power is calculated by the wattage meter, and the distance and temperature of the infrared lamp are measured. Finally, the appropriate temperature and distance of the infrared lamp to the human skin are estimated through calculation.

Keywords: Infrared, Far- infrared, Burn

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults over the age of 20 are not excluded from patients with lower back pain.

Exclusion Criteria:

1. Exclude cardiovascular diseases, anemia, high blood pressure and other diseases that may affect circulation.
2. People with skin diseases, skin allergies, and skin abnormalities.
3. Patients who are clinically diagnosed with cancer or other major injuries.
4. Excluded conditions are alcoholics, diabetic patients (blood sugar greater than or equal to 200 mg/dL), and severe or life-threatening complications (determined by the trial host based on medical history).
5. Women who are pregnant or breastfeeding (positive urine pregnancy test).
6. The moderator decides that it is not suitable to participate in this research.

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment of the Department of Traditional Chinese Medicine, Tainan Hospital, Ministry of Health and Welfare
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Body temperature of skin surface | 15 minutes
  Local body temperature of skin surface

SECONDARY OUTCOMES:
Distance from IR lamp to skin | 15 minutes
  IR lamp to skin

CONTACTS AND LOCATIONS:
Locations (1):
- Tainan Hospital, Ministry of Health and Welfare, Tainan, West Central Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided